CLINICAL TRIAL: NCT00443222
Title: An Open Trial With TNF Blockade With Infliximab (Remicade®), in Patients With Chronic Inflammatory Myopathies
Brief Title: Treatment With TNF Blockade, Infliximab, in Patients With Myositis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Schering-Plough (Industry); Medical Research Council (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Remicade myositis
Record Dates: First submitted 2007-03-02; First posted 2007-03-05 (Estimated); Last update posted 2007-03-05 (Estimated); Status verified 2007-03

CONDITIONS: Refractory Myositis
Keywords: infliximab; polymyositis; dermatomyositis; inclusion body myositis
MeSH Terms: conditions — Myositis; Polymyositis; Dermatomyositis; Myositis, Inclusion Body | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Infliximab

SUMMARY:
This is a 4 month open trial with TNF-blockade using infliximab (an antibody that blocks TNF) in adult patients with chronic myositis (polymyositis, dermatomyositis, inclusion body myositis) who have persisting muscle weakness and inflammatory active disease despite adequate treatment with immunosuppressives either currently or previously.

Infliximab is given as infusions, 5 mg/kg body weight, these infusions are repeated after 2, 6 and 14 weeks. The study involves 15 adult patients.

Primary outcome measure is muscle function assessed by muscle function index score.

Other outcome measures are Myositis Disease Activity core set: Patient's global assessment and physicians global assessment on visual analogue scales (VAS). Manual muscle test, Health assessment questionnaire (HAQ), serum levels of CPK, LD and extra muscular disease activity score. Muscle biopsy, Magnetic resonance imaging (MRI) of thigh muscles and Health related Quality of life, measured by SF-36.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients.
* Persisting muscle weakness defined as ≤ 80% of muscle strength as measured by functional index of myositis
* Signs of disease activity defined as muscle edema observed by magnetic resonance imaging (MRI) or creatine kinase (CK) elevation, or inflammatory cell infiltrates on muscle biopsy, and failure to respond to treatment with glucocorticoids for a minimum of six months in combination with azathioprine or methotrexate.

Exclusion Criteria:

* Pregnant women, nursing mothers or a planned pregnancy within one and a half years of enrolment.
* Prior administration of infliximab or any other therapeutic agent targeted at reducing TNF (e.g., Etanercept, pentoxifylline, thalidomide or anti-CD4+ antibody) within the previous six months.
* A history of known allergies to murine proteins.
* Serious infections, such as hepatitis, pneumonia, pyelonephritis in the previous 3 months. Less serious infections in the previous 3 months, such as acute upper respiratory tract infection (colds) or uncomplicated urinary tract infection (colds) or uncomplicated urinary tract infection need not to considered exclusions at the discretion of the treating physician.
* History of opportunistic infections such as herpes zoster within 2 months of screening. Evidence of active CMV, active pneumocystis carinii, drug resistant atypical mycobacterium, etc.
* Documented HIV infection.
* Current signs or symptoms of severe, progressive or uncontrolled renal, hepatic, hematologic, endocrine, pulmonary, cardiac, neurologic or cerebral disease.
* Any currently known malignancy or pre-malignant lesions or any history of malignancy within the past five years.
* Patients with alcoholism, alcoholic liver disease, or other chronic liver disease.
* Patients with a positive PPD and chest X-Ray suggestive of active TB or a previous exposure to TB.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid E Lundberg, MD, PhD, Principal Investigator — Rheumatology Unit, Department of Medicine, Karolinska University Hospital, Solna, Karolinska Institutet, Stockholm, Sweden